CLINICAL TRIAL: NCT05311670
Title: Pre-Implementation Study of Improving Thoracic Surgical Care Using Electronic Patient-Reported Outcomes (ePROS)
Acronym: TSPRO2
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC 2202; 1K23HL157765-01A1 (NIH)
Record Dates: First submitted 2022-03-10; First posted 2022-04-05 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Thoracic Surgery
Keywords: Electronic Patient-Reported Outcome
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-arm: Participants will be assigned to the single-arm involving monitoring of their symptoms.
  Interventions: Behavioral: Patient-reported outcomes monitoring

INTERVENTIONS:
Behavioral: Patient-reported outcomes monitoring — o Patient-reported outcomes will be collected from patients through web or telephone and alerts sent to providers.
  Other Names: Survey

SUMMARY:
The purpose of the LCCC 2202 is to evaluate the barriers and facilitators to implementing perioperative "ePRO monitoring". This study will inform a future hybrid effectiveness study (LCCC 2141:Improving Thoracic Surgical Care Using Electronic Patient-Reported Outcomes (ePROS). Eligible thoracic surgery patients will be enrolled to ePRO monitoring using web-based or telephone surveys. Patients will be asked to self-report symptoms for remote monitoring by their care team. Patients will be approached for a semi-structured interview to understand the barriers and facilitators to ePRO use.

DETAILED DESCRIPTION:
This is a single-site, non-randomized study in patients receiving major thoracic surgery, which commonly involves chest wall incisions and overnight admission Eligible patients will be approached at any time point between their preoperative clinic visit and up to 30 days after discharge from the hospital. Approximately 60 patients will be enrolled in the study. Patients will complete symptom surveys via email or telephone. Concerning symptoms will generate alerts for the clinical care team who will follow their usual protocols for the management of symptoms. Patients will be purposively selected and invited to participate in a semi-structured interview to understand their experience using ePRO. Interviews will continue until 30 complete interviews are obtained and/or thematic saturation is reached.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English speaking
* Able and willing to complete a web-based or telephonic symptom survey
* Planned to undergo surgery within 90 days or have undergone and been discharged from major thoracic surgery within the last 30 days.

Exclusion Criteria:

* Not completing planned surgery within 3 months of obtaining informed consent (for subjects recruited preoperatively)
* Inability to read and speak English
* Planned for foregut surgery (e.g. paraesophageal hernia repair, esophageal resection or repair)
* Having undergone only minor thoracic surgery (e.g. bronchoscopy, cervical mediastinoscopy)
* Dementia, altered mental status, or any psychiatric condition as determined by thoracic surgery provider team that would prohibit the understanding or rendering of informed consent.
* Current incarceration
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects scheduled thoracic surgery at UNC Chapel Hill Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Barriers to use of ePROs among patients | Up to one year (From one month after the study start until the thematic saturation is reached)
  Semi-structured interview with patients to evaluate ePRO use.
Facilitators to use of ePROs among patients | Up to one year (From one month after the study start until the thematic saturation is reached)
  Semi-structured interview with patients to evaluate ePRO use.

CONTACTS AND LOCATIONS:
Overall Officials: Gita Mody, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plan as of now to make IPD available to other researchers.

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials